CLINICAL TRIAL: NCT07244731
Title: Prognostic Evaluation of Red Blood Cell Distribution Width (RDW) in Severe and Critical COVID-19 Patients Monitored in the Intensive Care Unit
Brief Title: The Prognostic Role of Red Blood Cell Distribution (RDW) in Severe COVID-19 Patients
Acronym: RDW-Covıd-19
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice Güneş Yeşilova, MD, Specialist in Anesthesiology, Ankara University
Other Study IDs: HTCGNSTEZ; İ10-808-24 (Other: Ankara University Human Research Ethics Committee)
Record Dates: First submitted 2025-10-01; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: COVID - 19; Prognosis; ICU
Keywords: COVID-19; Red Cell Distribution Width (RDW); Mortality; Intubation; Prognostic marker
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to evaluate the prognostic significance of erythrocyte distribution width (RDW) in severe and critically ill COVID-19 patients followed in the intensive care unit (ICU). RDW is a parameter that measures the heterogeneity in red blood cell size and is associated with the pathophysiological processes of COVID-19, such as systemic inflammation, oxidative stress, and erythropoiesis disorders. This study investigated the relationship between RDW and the need for intubation and mortality, and its utility as a prognostic marker in COVID-19 patients.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is an infectious disease caused by the SARS-CoV-2 virus. According to official figures from the World Health Organization, the COVID-19 pandemic has sickened 780 million people worldwide and caused more than 7 million deaths.

Common symptoms of COVID-19 include fever, cough, and shortness of breath. Symptoms such as headache, sore throat, runny nose, muscle and joint pain, extreme fatigue, new-onset loss of smell and taste, and diarrhea may also occur. While the disease can be asymptomatic, severe cases can develop pneumonia, severe acute respiratory infection, multiple organ failure, and death. Predicting high risk in patients with COVID-19 has the potential to reduce mortality and morbidity by enabling early transfer of patients to intensive care units and planning appropriate treatment. For this purpose, numerous studies have been conducted to determine whether different markers can be used in addition to risk scores such as APACHE and SOFA, which are currently used in intensive care units. These markers include increased neutrophil and platelet counts, decreased lymphocyte counts, and elevated levels of B-type natriuretic peptide (BNP), blood urea nitrogen (BUN), creatine kinase (CK), bilirubin, interleukin-6 (IL-6), c-reactive protein (CRP), procalcitonin, ferritin, alanine aminotransferase (ALT), albumin, and lactate dehydrogenase (LDH). RDW (red blood cell distribution width), a measure of variation in red blood cell size, has traditionally been used in the diagnosis of various hematological conditions. In recent years, it has also been shown to be a potential marker of inflammation.

Increased proinflammatory activity and hypoxia impair erythropoiesis, leading to an increase in red cell distribution width (RDW) and changes in hematocrit. Increased RDW has been associated with poor prognosis in other critical illnesses, such as sepsis and cardiovascular disease. In COVID-19, viral inflammation can affect erythrocyte production and turnover, leading to an increase in RDW. Increased RDW increases proportionally with the degree of systemic inflammation and can therefore be a marker of disease severity. Higher RDW values at hospitalization have been associated with increased mortality and the need for intensive care. A meta-analysis of multiple studies has shown that high RDW is a strong predictor of mortality in COVID-19 patients. This meta-analysis suggests that RDW can be used as an early warning indicator to identify patients at high risk for severe disease and adverse clinical outcomes. Other research supports the use of RDW as a biomarker in COVID-19 and reinforces the role of RDW as a general marker of physiological stress/disease severity. RDW, a low-cost parameter included in the standard complete blood count, can be easily integrated into clinical practice, contributing to the early identification of high-risk COVID-19 patients and facilitating the planning of timely and appropriate medical interventions.

The aim of this study is to investigate the relationship between RDW values at admission and the need for intubation in severely ill and critically ill patients admitted to COVID-19 intensive care unit by analyzing the time course of RDW. Furthermore, the relationship between RDW and other laboratory and clinical parameters will also be investigated.

Materials and Methods: This retrospective study was conducted using data from patients admitted to the COVID-19 intensive care unit at Ankara University Ibn-i Sina Research and Application Hospital between April 2021 and August 2024. Among 758 patients admitted to the intensive care unit (ICU) due to COVID-19 between the specified dates and who met the World Health Organization's severe and critically ill COVID-19 criteria, 360 patients were randomly selected.

Patients' demographic characteristics (age, gender, vaccination status), comorbidities, length of stay in the ICU, need for intubation, laboratory parameters (RDW, hemoglobin, platelet count, leukocyte count, neutrophil/lymphocyte (N/L) ratio, CRP, procalcitonin, interleukin-6, etc.), and ICU severity scores (APACHE II and SOFA) were recorded. RDW values were recorded for five consecutive days, starting from the first day of ICU admission.

For statistical analyses, the Mann-Whitney U test was used to compare two independent groups, the Chi-square test for categorical variables, and the Two-Way Repeated Measurement ANOVA for repeated measurements. A P value of <0.05 was considered statistically significant. The prognostic value of RDW and the optimal cut-off value were determined using ROC analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Severe and critically ill COVID-19 patients (PCR test positivity of COVID)
* Patients who have been monitored in the intensive care unit for at least 3 days
* Patients without haematological malignancies

Exclusion Criteria:

* Patients under 18 years of age
* Those with haematological malignancies (as this may affect RDW levels)
* Patients who died within 3 days of admission to intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ministry of Health of the Republic of Turkey Ankara University Ibn-i-Sina Hospital Anaesthesiology and Resuscitation Department Patients admitted to the COVID-19 intensive care unit
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
discharge / death | From admission to the intensive care unit until ICU discharge or death, assessed up to 30 days.
  discharge from the intensive care unit / death during intensive care follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Necmettin Ünal, Study Director — Ankara University
Locations (1):
- Ankara University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT07244731/Prot_SAP_ICF_000.pdf